CLINICAL TRIAL: NCT01203826
Title: Extension Study of Protocol ENB-006-09 Evaluating the Long-term Safety and Efficacy of Asfotase Alfa (Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein) in Children With Hypophosphatasia (HPP)
Brief Title: Extension Study of Protocol ENB-006-09 - Study of Asfotase Alfa in Children With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-008-10
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- asfotase alfa (Experimental): asfotase alfa starting dose 3 mg/kg/week SC injection, increased to 6 mg/kg/week SC injection
  Interventions: Biological: Asfotase Alfa

INTERVENTIONS:
Biological: Asfotase Alfa
  Other Names: human recombinant tissue nonspecific alkaline phosphatase fusion protein

SUMMARY:
This clinical trial studies the long term safety and efficacy of asfotase alfa in children with HPP who completed Study ENB-006-09 (NCT00952484).

DETAILED DESCRIPTION:
Asfotase alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

* Compliant and satisfactory completion of Enobia-sponsored clinical trial ENB-006-09
* Written informed consent by parent or other legal guardian prior to any study procedures being performed
* Parent or other legal guardian willing to comply with study requirements

Exclusion Criteria:

* Clinically significant disease that precludes study participation, in the Investigator's opinion
* Treatment with an investigational drug other than asfotase alfa
* Enrollment in any study (other than ENB-006-09) involving an investigational drug, device, or treatment for HPP
* Prior treatment with bisphosphonates

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Shriners Hospital for Children, St Louis, Missouri, United States
- Children's Hospital Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Simmons JH, Rush ET, Petryk A, Zhou S, Martos-Moreno GA. Dual X-ray absorptiometry has limited utility in detecting bone pathology in children with hypophosphatasia: A pooled post hoc analysis of asfotase alfa clinical trial data. Bone. 2020 Aug;137:115413. doi: 10.1016/j.bone.2020.115413. Epub 2020 May 14. PMID 32417537
- [Derived] Whyte MP, Madson KL, Phillips D, Reeves AL, McAlister WH, Yakimoski A, Mack KE, Hamilton K, Kagan K, Fujita KP, Thompson DD, Moseley S, Odrljin T, Rockman-Greenberg C. Asfotase alfa therapy for children with hypophosphatasia. JCI Insight. 2016 Jun 16;1(9):e85971. doi: 10.1172/jci.insight.85971. PMID 27699270
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main criteria for inclusion in Study ENB-006-09 were patients ages 5 to 12 years inclusive, with open growth plates at time of study entry and a documented diagnosis of HPP. To enter the extension, Study ENB-008-10, patients had to successfully complete Study ENB-006-09 and provide consent.
Groups:
- 2 mg/kg Asfotase Alfa; 3 mg/kg Asfotase Alfa: The starting dose of asfotase alfa was 3 mg/kg/week for all patients in Study ENB-008-10 and was subsequently increased per study-wide dose adjustment to a total dose of 6 mg/kg/week. Results are shown by the patient's dose group assignment from Study ENB-006-09.
Period: Overall Study
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Started | 6 (Dose cohorts are per assigned dose in ENB-006-09. Results presented are for Study ENB-008-10 only.) | 6 (Dose cohorts are per assigned dose in ENB-006-09. Results presented are for Study ENB-008-10 only.)
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 mg/kg Asfotase Alfa; 3 mg/kg Asfotase Alfa: Dose group shown is as per patient's randomization in Study ENB-006-09
- Total: Total of all reporting groups
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Enrollment
  years | 8.4 (2.21) | 9.0 (2.51) | 8.7 (2.27)
Age, Customized [Count of Participants; unit: Participants] — n %
  Participants
    Age Group at Enrollment: 2 to 11 Years; % | 5 | 5 | 10
    Age Group at Enrollment: 12 to 17 Years; % | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — n %
  Participants
    Female | 1 | 1 | 2
    Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — n %
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 5 | 6 | 11
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — n %
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 6 | 6 | 12
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 1 | 3
  United States | 4 | 5 | 9
Hypophosphatasia Phenotype [Count of Participants; unit: Participants] — n %
  Participants
    Infantile (< 6 months) | 3 | 1 | 4
    Juvenile (≥ 6 months to < 18 yrs) | 3 | 5 | 8
Age at Onset of Hypophosphatasia Symptoms [Mean (Standard Deviation); unit: Months] | 10.8 (8.66) | 11.5 (5.54) | 11.2 (6.94)
Tanner Stage 1 [Count of Participants; unit: Participants] — n %; Tanner Stage 1 = Prepubertal children
  Participants | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Radiograph Evaluation Using a Qualitative Radiographic Global Impression of Change (RGI-C) Scale Compared to Baseline (Pre-treatment) in Study ENB-006-09.
Description: Evaluation of radiographic change in rickets severity (as assessed by skeletal radiographs of the hands/wrists and knees) from the Baseline of Study ENB-006-09 (NCT00952484) to the End of Study (EOS) visit in Study ENB-008-10 using an ordinal RGI-C scale score. The RGI-C is a 7-point rating scale that ranges from -3 (indicative of severe worsening of HPP associated rickets) to +3 (indicative of complete or near complete healing of HPP associated rickets).
  The time points will be pre-treatment (Baseline from Study ENB-006-09) to the last radiographic assessment in Study ENB-008-10, which represents at least 72 months of treatment.
Time Frame: At least 72 months of treatment with asfotase alfa
Population: Each visit in Study ENB-008-10 was calculated relative to the start of exposure to asfotase alfa in Study ENB-006-09 (NCT00952484); 24 weeks are added to each visit in Study ENB-008-10. Results shown are for the last assessment in Study ENB-008-10 and represent at least 72 months of treatment with asfotase alfa.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Asfotase Alfa Combined: ITT population for Study ENB-008-10, which included all patients that received treatment with asfotase alfa.
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
units on a scale | 2.83 [2.0 to 3.0]
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Change is relative to Baseline in Study ENB-006-09 (NCT00952484). The RGI-C score represents evaluations of skeletal X-rays at each post-treatment study timepoint in Study ENB-008-10 compared with pre-treatment X-rays from Study ENB-006-09, using an ordinal scale. Therefore, no Baseline data for RGI-C are available; Test type: Other; p = 0.0005, Wilcoxon signed-rank test; P-value based on Wilcoxon signed-rank test

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs are events starting on or after the day of first dose of asfotase alfa and recorded in Study ENB-008-10 (at least 66 months of treatment in Study ENB-008-10).
Groups:
- Combined Asfotase Alfa Group: All patients treated with asfotase alfa during Study ENB-008-10
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa | Combined Asfotase Alfa Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/kg Asfotase Alfa (N=6) | 3 mg/kg Asfotase Alfa (N=6) | Combined Asfotase Alfa Group (N=12)
Injection site erythema (General disorders) | 4 (18) | 6 (27) | 10 (45)
Injection site macule (General disorders) | 4 (28) | 5 (31) | 9 (59)
Injection site hypertrophy (General disorders) | 4 (14) | 4 (13) | 8 (27)
Injection site atrophy (General disorders) | 3 (10) | 3 (8) | 6 (18)
Injection site discolouration (General disorders) | 2 (8) | 2 (8) | 4 (16)
Fatigue (General disorders) | 1 (2) | 2 (2) | 3 (4)
Gait disturbance (General disorders) | 0 (0) | 3 (3) | 3 (3)
Injection site pain (General disorders) | 2 (6) | 1 (2) | 3 (8)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3)
Injection site pruritis (General disorders) | 2 (12) | 0 (0) | 2 (12)
Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site papule (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (7) | 1 (7)
Upper respiratory tract infection (Infections and infestations) | 5 (24) | 4 (20) | 9 (44)
Gastroenteritis (Infections and infestations) | 2 (3) | 3 (5) | 5 (8)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (2) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 3 (3)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (3)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (2) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 3 (6)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Epiphyses premature fusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (3)
Oral pain (Gastrointestinal disorders) | 1 (3) | 1 (1) | 2 (4)
Dental discomfort (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tooth crowding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival deposit (Eye disorders) | 3 (5) | 3 (3) | 6 (8)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Corneal deposits (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Optic atrophy (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Optic disc drusen (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Retinal vascular disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (15) | 3 (4) | 6 (19)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (7) | 0 (0) | 1 (7)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (7) | 1 (1) | 3 (8)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 1 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (6) | 2 (6)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Growth hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less